CLINICAL TRIAL: NCT05515211
Title: Diagnostic Accuracy of Foot Length in Predicting Preterm and Low Birth Weight Using Ultrasound Dating as The Gold Standard in a Rural District of Pakistan
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Shiyam Sunder, MBBS, MSc, Assistant Professor, Aga Khan University
Other Study IDs: 2022-7421-21580
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Preterm Birth; Low Birth Weight
Keywords: Gestational age; birth weight; Diagnostic accuracy; Regression equation; Correlation
MeSH Terms: conditions — Premature Birth; Birth Weight

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Foot length — Foot length will be measured from the midpoint of the heel to the longest toe.

SUMMARY:
Background:

The burden of preterm and low birth weight babies (LBW) is high in low- and middle-income countries (LMICs). Therefore, assessment of gestational age (GA) and birth weight is important. The GA is assessed using a reliable last menstrual period (LMP), measuring fundal height, using ultrasound for dating, or postnatally using Ballard, Dubowitz, or Eregie scores. However, each method has some limitations. Pregnant women in LMIC are not able to recall LMP and are also unreliable when menstrual cycles are irregular, fundal height is often imprecise and subject to variation due to observer bias, uterine pathologies, abdominal obesity, amniotic fluid volume, fetal position, and ultrasound in a rural setting is often unreliable because lack of trained sonologist, power failures, and maintenance of ultrasound machine. Post-natal GA scoring is also lengthy, subjective, and time-consuming. Similarly, determining birth weight has many challenges. In Thatta, weighing scales are only available in health facilities, therefore, birth weight is available for babies born in the health facilities. Furthermore, even where weighing scales are available, the calibration and maintenance are not without challenges, especially in the extremely hot climate. In the majority of studies, foot length has been validated for determining GA and birth weight, with LMP serving as the gold standard, which has limitations in our population. In a meta-analysis on the diagnostic accuracy of foot length to identify preterm and LBW, researchers emphasized the need for studies using high-quality ultrasound as a reference standard for early dating. Hence, there is a need to develop a simple and effective method of GA and birth weight that healthcare providers of all levels including mid-level healthcare workers in remote areas can use with reasonable accuracy.

Objectives of the study The primary objectives of the study are to determine the diagnostic accuracy of foot length in predicting GA and low birth weight using ultrasound conducted between 6-20 weeks for the predicted estimated date of delivery (EDD) as the gold standard.

Secondary objectives of the study are, 1) to develop the regression equations that predict gestational age and low birth weight using foot length, 2) to assess the use of foot length measurement as a screening tool to identify LBW or preterm infants in a community-based setting, and 3) to develop percentile charts of foot length for gestational age and low birth weight

Methods:

This test validation study will be conducted in Global Network's Maternal and Newborn Health Registry catchment area. All live birth singleton babies who have a first-trimester ultrasound for gestational age and birth weight within 48 hours of birth will be included in this study. Stillbirths, multiple pregnancies, gross congenital malformations such as neural tube defects, omphalocele, etc., club foot, and babies with chromosomal abnormalities such as Down syndrome that make measuring foot length difficult, will be excluded from the study. Gestational age will be assessed using ultrasound between 6-20 weeks of gestation by a trained sonographer working in the registry. Neonatal assessment having neuromuscular, and physical signs will be conducted by the research assistants (RA). RA will be taking anthropometric measurements such as birth weight using calibrated weighing scales, foot length, mid-upper arm circumference, and fronto-occipital circumference.

The data will be entered in Epicollect data five. Sensitivity, specificity, positive & negative predictive value, likelihood ratios, and diagnostic accuracy will be done using different cut-offs of foot length against ultrasound estimated gestational age and birth weight. Receivers operating characteristics (ROC) curves will be generated to identify the optimal cut-off point for foot length taken within 24 hours of birth for identification of prematurity and LBW (based on first-trimester ultrasound) with ≥80% sensitivity. Linear regression will be done for estimating predictive values of foot length by GA. Pentile charts for foot length (FL) against GA will be derived. Bland Altman's analyses will identify and quantify any biases inherent to the tool.

Public health implications:

If these equations predict gestational age and birth weight with accuracy, an android-based application can be developed for health care providers (HCP) who simply measure foot length and enter it into the application to identify preterm &/or low birth weight along with referred guidelines for early treatment. This is one step closer to Every Newborn Action Plan's goal of lowering neonatal mortality to 12/1000 LB by 2030.

ELIGIBILITY:
Inclusion Criteria:

* All livebirth singleton babies
* Having first-trimester ultrasound for gestational age
* Birth weight measured within 48 hours of birth

Exclusion Criteria:

* Stillbirths
* Multiple pregnancies
* Gross congenital malformations such as neural tube defects, omphalocele, etc.,
* Club foot
* Pregnant women whose ultrasound dating differs between sonographers and senior radiologists

Ages: 0 Hours to 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Singleton alive newborns
Sampling Method: Non-Probability Sample
Enrollment: 336 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-13 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of foot length for preterm baby | Within 48 hours of birth
  Diagnostic accuracy defined as sensitivity, specificity, predictive values, likelihood ratios
Diagnostic accuracy of foot length for low birth weight baby | Within 48 hours of birth
  Diagnostic accuracy defined as sensitivity, specificity, predictive values, likelihood ratios

SECONDARY OUTCOMES:
Small for gestational age | Within 48 hours of birth
  Birth weigh less than 10th centile for age and sex

CONTACTS AND LOCATIONS:
Locations (1):
- Community of Thatta, Thatta, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
After the publication of the main papers, data could be made publicly available to other researchers.

REFERENCES:
- [Derived] Tikmani SS, Brown N, Inayat Ali A, Martensson A, Saleem S, Martensson T. Postnatal foot length measurement as a proxy to identify low birth weight for frontline health workers in rural Sindh Province, Pakistan: a diagnostic accuracy study. BMJ Open. 2024 Dec 26;14(12):e089153. doi: 10.1136/bmjopen-2024-089153. PMID 39730154
- [Derived] Tikmani SS, Brown N, Inayat A, Martensson A, Saleem S, Martensson T. Diagnostic accuracy of foot length measurement for identification of preterm newborn in rural Sindh, Pakistan. BMJ Paediatr Open. 2024 Jan 24;8(1):e002316. doi: 10.1136/bmjpo-2023-002316. PMID 38267220